CLINICAL TRIAL: NCT05392803
Title: Pulsed Electromagnetic Fields for Post-Amputation Pain: A Randomized, Triple-Masked, Sham-Controlled, Crossover Pilot Study
Brief Title: Pulsed Electromagnetic Fields for Post-Amputation Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PEMF Amputee Pilot
Record Dates: First submitted 2022-05-19; First posted 2022-05-26 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Phantom Limb Pain; Residual Limb Pain
MeSH Terms: conditions — Phantom Limb | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either active or sham treatment for 30 days; and will then crossover and receive the alternative treatment for 30 additional days. The primary analysis will compare the initially-randomized active and sham treatment groups--thus, a parallel group (inter-participant) comparison; but secondary analyses will compare intra-participant changes as well.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Drug Service will create the randomization tables and provide the investigators with the appropriate device (active or sham), leaving all participants, investigators, and the statistician masked to treatment group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active then Sham Treatment (Experimental): Application of 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy, 7 day "washout", 30 days of sham.
  Interventions: Device: Active then Sham Treatment
- Sham then Active Treatment (Experimental): Application of 30 days of a nonfunctional sham device, 7 day "washout", then 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy
  Interventions: Device: Sham then Active Treatment

INTERVENTIONS:
Device: Active then Sham Treatment — Application of 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy; then sham treatment after a 7-day "washout" period
  Other Names: nonthermal, pulsed shortwave (radiofrequency) therapy then sham; pulsed electromagnetic fields therapy then sham
  Arms: Active then Sham Treatment
Device: Sham then Active Treatment — Application of 30 days of sham treatment; then 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy after a 7-day "washout" period
  Other Names: Sham then nonthermal, pulsed shortwave (radiofrequency) therapy; Sham then pulsed electromagnetic fields therapy
  Arms: Sham then Active Treatment

SUMMARY:
Pulsed electromagnetic field therapy is a possible method of pain control involving the application of electromagnetic energy (also termed nonthermal, pulsed, shortwave radiofrequency therapy). Food and Drug Administration-cleared devices have been in clinical use for over 70 years. For decades, available devices consisted of a large signal generator and bulky coil applicator that were not portable and produced significant electromagnetic interference, making them impractical for common use. However, small, lightweight, relatively inexpensive, noninvasive, Food and Drug Administration-cleared devices that function for 30 days are now available to treat acute and chronic pain, decrease inflammation and edema, and hasten wound healing and bone regeneration. Therefore, it has the potential to concurrently improve analgesia and decrease or even negate opioid requirements, only without the limitations of opioids and peripheral nerve blocks. The purpose of this pilot study is to explore the possibility of treating chronic post-amputation pain with nonthermal, pulsed shortwave (radiofrequency) therapy, optimize the study protocol, and estimate the treatment effect in preparation for developing subsequent definitive clinical trials.

DETAILED DESCRIPTION:
The proposed study will be a randomized, participant- and observer-masked, sham-controlled, crossover, human participants pilot study with two primary aims:

Specific Aim 1: To determine the feasibility and optimize the protocol for subsequent clinical trials that will compare the addition of nonthermal, pulsed shortwave therapy to usual and customary analgesia for post-amputation phantom and residual limb pain.

Specific Aim 2: To estimate the treatment effect of adding nonthermal, pulsed shortwave therapy to usual and customary analgesia for post-amputation phantom and residual limb pain. This will provide an idea of the optimal amputee characteristics amenable to this analgesic technique and allow determination of the required sample sizes of subsequent definitive clinical trials.

Hypothesis: Nonthermal, pulsed shortwave therapy will decrease pain in the 28 days following application for post-amputation pain.

This will be a single-center (University of California San Diego), randomized, participant- and observer-masked, sham-controlled, crossover human subjects pilot study.

Enrollment. Participants will be consenting adults experiencing post-amputation phantom and/or residual limb pain. Study inclusion will be proposed after an amputee contacts the investigators. If an individual desires study participation, written, informed consent will be obtained using a current University of California San Diego Institutional Review Board-approved informed consent form. The study population of interest includes adult women and men of all races, ethnicity, sexual identity, and socioeconomic status.

Procedures. Following written, informed consent, we will record baseline anthropometric information (age, sex, height, weight, amputation details and current pain levels).

Treatment Group Assignment. Each participant will be randomized to one of two treatment groups: Active or Sham treatment. There are sham devices produced that are identical to active devices, only they do not deliver pulsed electromagnetic energy. Randomization will be in block sizes of 2. The computer-generated randomization lists will be created by the University of California San Diego Investigational Drug Service in a 1:1 treatment group ratio using opaque envelopes. The active and sham devices are indistinguishable in appearance, and therefore investigators, participants, and all clinical staff other than the individual who opens the randomization envelope and chooses a sham or active device will be masked to treatment group assignment for the duration of the data collection period. An Investigational Drug Service pharmacist will open the envelope and provide the investigators with the appropriate device, keeping all investigators masked to treatment group assignment. Upon completion of data collection, the pharmacist will provide the investigators with a masked list of the treatment groups (e.g., "Treatment A" and "Treatment B"), and the active/sham lists only following analysis for that subgroup, resulting in a triple-masked study (investigators, participants, statistician).

Study intervention. The pulsed shortwave devices used are over-the-counter (Model 088, BioElectronics, Frederick, Maryland) and 2 devices (both the same treatment group) will be shipped to the patient either in or out of California who will then contact an investigator for assistance in self-placement of the device on the residual limb. The optimal location to treat phantom pain is currently unknown and will partially informed by the results of this pilot study, and patients will be encouraged to move the devices to a new anatomic location every two days until relief is experienced.

Supplemental analgesics. In addition to the pulsed shortwave device(s), participants will receive standard-of-care supplemental analgesics which can include acetaminophen, ibuprofen, ketorolac, opioids, gabapentin (this is provider- and patient-dependent). Therefore, all patients of this study-regardless of the treatment arm they are randomized to-will continue to receive current usual and customary analgesia: all will receive the same combination of supplemental analgesics they would regardless of study participation. Participants will be provided with verbal and written instructions, and the telephone and pager numbers of an investigator available during business hours throughout the treatment period. Participants can shower with the device in place, but not submerge it during swimming or a bath, as advised by the manufacturer.

Amputees will return their initial devices in pre-addressed and -stamped envelopes that we provide. They will be sent a second device which is the opposite treatment of the initial device: participants who initially received sham will subsequently receive active, and vice versa. These will be applied on (approximately) Day 35 and the same protocol will be repeated as for the initial device, with additional data collected for 35 days after placement of the second device. The second device will be discarded in the trash.

Of note, if a device is reported lost or nonfunctional during the study, it will be replaced by the investigators by mail if more than 7 days of treatment remain.

Primary end points: This is an exploratory pilot study to assist in planning subsequent definitive trials and we therefore have no data analysis plan. We will enroll a convenience sample of up to 40 participants. The outcome measures of primary interest will be (1) the change in "average" residual and phantom limb pain scores between baseline and Day 28 of the initial treatment, as well as (2) the Patient Global Impression of Change on Day 28 of the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult patients of at least 18 years of age [19 years in Alabama and Nebraska]
* with an upper or lower limb amputation at least 12 weeks prior to enrollment distal to the shoulder or hip (femoral head remaining), respectively, and including at least one metacarpal or metatarsal bone, respectively
* experience at least moderate residual and/or phantom limb pain-defined as a 3 or higher on the Numeric Rating Scale (NRS; 0-10, 0= no pain; 10=worst imaginable pain)-at least daily for the previous 2 months
* willing to avoid both changes to their analgesic regimen as well as elective surgical procedures for 70 days after initiation of treatment with PEMF therapy

Exclusion Criteria:

* concurrent use of an implanted pulse generator (e.g., cardiac pacemaker)
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- Univerity of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Intervention (30 Days), Washout (7 Days), Sham Intervention (30 Days): Application of 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy, 7 day "washout", 30 days of sham intervention.
- Sham Intervention (30 Days), Washout (7 Days), Active Intervention (30 Days): Application of 30 days of a nonfunctional sham device, 7 day "washout", then 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy
Period: Overall Study
Arm/Group | Active Intervention (30 Days), Washout (7 Days), Sham Intervention (30 Days) | Sham Intervention (30 Days), Washout (7 Days), Active Intervention (30 Days)
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Then Sham Treatment | Sham Then Active Treatment | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (14) | 61 (22) | 59 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 3 | 5 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 7 | 14
Height [Mean (Standard Deviation); unit: cm] | 180 (9) | 172 (9) | 176 (9)
Weight [Mean (Standard Deviation); unit: kg] | 84 (21) | 69 (18) | 76 (20)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26 (6) | 23 (4) | 24 (5)
Trans-Femoral amputation [Count of Participants; unit: Participants] | 3 | 7 | 10
Trans-Tibial amputation [Count of Participants; unit: Participants] | 4 | 0 | 4
Continuous phantom limb pain at baseline [Count of Participants; unit: Participants] | 6 | 5 | 11
Continuous residual limb pain at baseline [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Average RESIDUAL Limb Pain Scores Between Baseline and Day 28 of the Initial Treatment as Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will be the difference between the baseline and Day 28 timepoints.
Time Frame: Baseline and Day 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Active Treatment: Application of 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy
- Sham Treatment: Application of 30 days of a nonfunctional sham device
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale | 2.5 [2.5 to 2.8] | 0 [-0.5 to 0]

2. Primary Outcome: Change in Average PHANTOM Limb Pain Scores Between Baseline and Day 28 of the Initial Treatment as Measured With the Numeric Rating Scale
Description: as for outcome 1
Time Frame: Baseline and Day 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale | 2.3 [1.8 to 3.5] | 0 [-0.3 to 0]

3. Primary Outcome: Patient Global Impression of Change for RESIDUAL Limb Pain Between Baseline and Day 28 of the Initial Treatment
Description: A 7-point Likert scale with 1 equivalent to "much worse", 4 equivalent to "no change", and 7 equivalent to "much improved". Patients compare their current pain level with baseline using this scale.
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale | 7 [4 to 7] | 4 [4 to 4]

4. Primary Outcome: Patient Global Impression of Change for PHANTOM Limb Pain Between Baseline and Day 28 of the Initial Treatment
Description: as for outcome 3
Time Frame: Day 28
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale | 6.5 [4 to 7] | 4 [4 to 4]

5. Secondary Outcome: Patient Global Impression of Change for RESIDUAL Limb Pain
Description: as for outcome 3
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 2 | 4 [4 to 6] | 4 [4 to 5]
  Day 4 | 5 [4 to 7] | 4 [4 to 4]
  Day 7 | 5 [4 to 7] | 4 [4 to 4.5]
  Day 21 | 7 [4 to 7] | 4 [4 to 4]
  Day 28 | 7 [4 to 7] | 4 [4 to 4]
  Day 35 | 4 [4 to 7] | 4 [4 to 4]

6. Secondary Outcome: Patient Global Impression of Change for PHANTOM Limb Pain
Description: as for outcome 3
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 2 | 5 [4 to 7] | 4 [4 to 4]
  Day 4 | 5 [4 to 7] | 4 [3.5 to 4]
  Day 7 | 6.5 [4 to 7] | 4 [4 to 4.3]
  Day 21 | 6.5 [4 to 7] | 4 [4 to 4.5]
  Day 28 | 6.5 [4 to 7] | 4 [4 to 4]
  Day 35 | 4 [4 to 6] | 4 [4 to 4]

7. Secondary Outcome: Change in AVERAGE RESIDUAL Pain From Baseline Measured With the Numeric Rating Scale
Description: The numeric rating scale is a 0-10 Likert scale measuring pain level with 0 = no pain and 10 = worst imaginable pain scale. The outcome will the difference between the baseline and current pain level measured with the Numeric Rating Scale
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 2 | 2.5 [1.3 to 3.8] | 4 [2 to 5]
  Day 4 | 3 [1.4 to 3.8] | 4 [4 to 6]
  Day 7 | 2 [1 to 3.3] | 4 [4 to 4]
  Day 21 | 1.3 [0.8 to 3.1] | 4 [4 to 4.5]
  Day 28 | 1.5 [0.8 to 2.5] | 4 [4 to 4.5]
  Day 35 | 1.5 [1 to 4] | 4 [4 to 5.5]

8. Secondary Outcome: Change in WORST RESIDUAL Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 2 | 3.5 [3 to 5.5] | 5 [3 to 7]
  Day 4 | 3 [2.5 to 6.5] | 5 [5 to 9]
  Day 7 | 3 [2.3 to 5] | 5 [5 to 6]
  Day 21 | 3 [1.5 to 5] | 5.5 [5 to 7]
  Day 28 | 3 [1.5 to 5] | 5.5 [5 to 6.5]
  Day 35 | 4 [2.3 to 6.5] | 5 [4.5 to 7]

9. Secondary Outcome: Change in LEAST RESIDUAL Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 28 and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 28 | 0 [0 to 0] | 3.5 [0 to 6]
  Day 35 | 0 [0 to 0.5] | 0 [0 to 0.5]

10. Secondary Outcome: Change in CURRENT RESIDUAL Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 28 and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 28 | 0 [0 to 2] | 4 [3 to 4]
  Day 35 | 1 [0 to 2] | 1 [0 to 2]

11. Secondary Outcome: Change in AVERAGE PHANTOM Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
units on a scale
  Day 2 | 4.5 [1.5 to 5.8] | 3 [2.3 to 3.5]
  Day 4 | 4 [2.3 to 5] | 3.5 [3 to 4]
  Day 7 | 2 [1.1 to 5.6] | 4 [3.3 to 5.8]
  Day 21 | 2 [0 to 4.6] | 4 [3 to 5.3]
  Day 28 | 2 [0 to 4.3] | 4 [3.8 to 5.5]
  Day 35 | 2.5 [1.5 to 4.5] | 4 [3.9 to 4.8]

12. Secondary Outcome: Change in WORST PHANTOM Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 2, 4, 7, 21, 28, and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 2 | 6 [4.3 to 7] | 5 [3.8 to 7]
  Day 4 | 4.7 [1.8 to 7.4] | 6.5 [4.5 to 10]
  Day 7 | 3.5 [1.5 to 7.3] | 5 [4.5 to 7.8]
  Day 21 | 3.5 [1 to 5.1] | 5 [3 to 8.3]
  Day 28 | 3.5 [.9 to 7.3] | 6 [4.5 to 9.3]
  Day 35 | 5 [3.8 to 8] | 5.5 [4.8 to 7]

13. Secondary Outcome: Change in LEAST PHANTOM Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 28 and 35
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
units on a scale
  Day 28 | 0 [0 to 3.6] | 0 [0 to 1.5]
  Day 35 | 0 [0 to 3.7] | 1 [0 to 3.3]

14. Secondary Outcome: Change in CURRENT PHANTOM Pain From Baseline Measured With the Numeric Rating Scale
Description: as for outcome 7
Time Frame: Days 28 and 35
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 28 | 3 [1 to 4.5] | 3 [0 to 4]
  Day 35 | 3.5 [.8 to 4.8] | 4 [3 to 4.8]

15. Secondary Outcome: As-needed (Non-scheduled) Analgesic Use
Description: Patient's perception of requirements over the previous 24 hours of as-needed (non-scheduled) analgesic use
Time Frame: Inquired on Day 2, 4, 7, 21, 28 and 35 for both initial and crossover treatments
Population: This outcome was inadvertently left off the case report forms, and therefore no data was collected for this outcome
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Brief Pain Inventory, Short Form (Interference Sub Scale)
Description: The Brief pain Inventory (short form) is an instrument specifically designed to assess pain and its impact on physical and emotional functioning. The brief Inventory is comprised of three domains: (1) pain, with four questions involving "worst", "average" and "current" pain levels using a 0-10 numeric rating scale [we are not using]; (2) percentage of relief provided by pain treatments with one question [we are not using] and, (3) interference with 7 questions involving physical and emotional functioning using a 0-10 Likert scale [0=no interference (good); 10=complete interference (bad)]: general activity, mood, walking ability, normal work, relations with other people, sleep and enjoyment of life. This outcome will include the interference subscale: 0=no interference (good); 70=complete interference (bad)
Time Frame: Inquired on Days 28 and 35
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Day 28 | 19.7 (20.4) | 20.9 (5.2)
  Day 35 | 34 (26) | 28 (20)

17. Secondary Outcome: Awakenings Due to Pain the Previous Evening
Description: The number of awakenings due to pain that occurred the previous evening
Time Frame: Inquired on Days 2, 4, 7, 21, 28, and 35
Measure: Mean (Standard Deviation); unit: number of awakenings
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
number of awakenings
  Day 2 | 0 (0) | .1 (.4)
  Day 4 | .6 (.9) | 1.9 (3.7)
  Day 7 | .4 (.9) | .1 (.4)
  Day 21 | 0 (0) | .1 (.4)
  Day 28 | .4 (.9) | .3 (.8)
  Day 35 | .4 (.9) | 2.6 (3.7)

18. Secondary Outcome: Does Patient Want to Continue Using Device (Participants Answering "Yes")?
Description: Does the patient want to continue using device answered as "yes" or "no". "Yes" means they DO want to continue using the device, while "no" means they do NOT want to continue using the device.
Time Frame: Inquired on Day 35
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
Participants | 7 | 2

19. Secondary Outcome: Device Location Changes
Description: If a patient moves the anatomic location of one or both of the intervention devices (and where the device is moved to) since the last contact
Time Frame: Inquired on Days 2, 4, 7, 21, 28 and 35
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Sham Treatment
Number analyzed (Participants) | 12 | 14
Participants
  Day 2 | 0 | 0
  Day 4 | 1 | 0
  Day 7 | 1 | 0
  Day 21 | 0 | 0
  Day 28 | 0 | 0
  Day 35 | 0 | 0

ADVERSE EVENTS:
Time Frame: For participants who had only the initial treatment, the follow-up was 35 days. For participants who participated in both the initial and crossover treatments, the follow-up was 70 days.
Groups:
- Active: Application of 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy, 7 day "washout", 30 days of sham
- Sham: Application of 30 days of a nonfunctional sham device, 7 day "washout", then 30 days of nonthermal, pulsed shortwave (radiofrequency) therapy
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/14
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05392803/Prot_SAP_000.pdf